CLINICAL TRIAL: NCT01675375
Title: Laser Vision Correction Use of an Eye Shield for Maintaining Vision and Mitigating Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FORSIGHT Vision3 (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CS 004
Record Dates: First submitted 2012-08-28; First posted 2012-08-29 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Post Laser Vision Correction Pain and Discomfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eye shield (Experimental): Eye shield place on post Laser Vision Correction eye
  Interventions: Device: Eye Shield

INTERVENTIONS:
Device: Eye Shield — one application following refractive surgery

SUMMARY:
The purpose of this research is to determine if an investigational thin shield can effectively reduce discomfort following Laser Vision Correction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo Laser Vision Correction for correction of refractive error
* FDA approved treatment guidelines for Laser Vision Correction
* Age 18-60
* Patients able to understand the requirements of the study, willing to follow study instructions, provide written informed consent to participate, and comply with all study requirements, including the required study follow-up visits

Exclusion Criteria:

* Any other anterior segment abnormality other than that associated with LAser Vision Correction
* Any abnormalities associated with the eye lids
* Uncontrolled blepharitis or dry eye
* Prior laser treatment of the retina
* Any ophthalmic surgery performed within three (3) months prior to study excluding PRK or LASIK
* Diagnosis of glaucoma
* Active diabetic retinopathy
* Clinically significant inflammation or infection within six (6) months prior to study
* Uncontrolled systemic disease (e.g., diabetes, hypertension, etc.) in the opinion of the Investigator
* Participation in any study involving an investigational drug within the past 30 calendar days, or ongoing participation in a study with an investigational material
* Intolerance or hypersensitivity to topical anesthetics, antibiotics, steroids or any other pharmaceuticals that may be used pre and post surgically
* Specifically known intolerance or hypersensitivity to contact lenses or any component of the investigative material
* A medical condition, serious concurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up
* Any condition that, in the opinion of the investigator, would jeopardize the safety of the patient
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Evidence of maintaining vision and mitigating pain post Laser Vision Correction using an Eye Shield | 1yr
  Evidence of maintaining vision and mitigating pain post Laser Vision Correction using an Eye Shield by subjective patient questionnaires and objective imaging and slit lamp examination.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - ClearView Eye and Laser, San Diego, California
  - Kraff Eye Institute, Chicago, Illinois
  - Talamo Laser Eye Consultants, Boston, Massachusetts
  - Physicians Protocol, Greensboro, North Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota